CLINICAL TRIAL: NCT03321461
Title: Novel Tumor Targeted Fluorescent TMTP1-ICG Mapping in Colposcopy-directed Biopsy
Brief Title: TMTP1-ICG Mapping in Colposcopy-directed Biopsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Director, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TMTP1-ICG-02
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMTP1 (Experimental): The TMTP1-ICG (WuXi AppTec, Shanghai, China) powder was diluted in 20 ml of aqueous sterile water to a concentration of 1.0 mg/mL. Then TMTP1-ICG spray was applied thoroughly to the ectocervix for 30 minutes. After cleaned by NS, fluorescent detected sites will be removed.
  Interventions: Drug: TMTP1
- ICG (Active Comparator): The ICG (WuXi AppTec, Shanghai, China) powder was diluted in 20 ml of aqueous sterile water to a concentration of 1.0 mg/mL. ICG spray was applied thoroughly to the ectocervix for 30 minutes. After cleaned by NS, fluorescent detected sites will be removed.
  Interventions: Drug: ICG

INTERVENTIONS:
Drug: TMTP1 — Fluorescent sites will be removed
  Arms: TMTP1
Drug: ICG — Fluorescent sites will be removed
  Arms: ICG

SUMMARY:
Investigators aimed to determine the validity of the novel tumor targeted fluorescent TMTP1-ICG to increased accuracy of colposcopy-directed biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Suspicious of cervical disease required a colposcopy-directed biopsy.
* Subjects must sign an informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

* Breast-feeding or pregnant.
* Ongoing participation in another clinical trial with an investigational drug with 3 months.
* Own allergy towards ICG and/or alcohol.
* Diagnosis of bacterial vaginosis, fungal vaginitis, sexually transmitted diseases.
* Patients with cardiac dysfunction or hepatic insufficiency or renal insufficiency.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 day
  Sensitivity of fluorescent detection of TMTP1-ICG compared to the sensitivity of ICG

SECONDARY OUTCOMES:
Specificity | 7 days
  Specificity of fluorescent detection of TMTP1-ICG compared to the sensitivity of ICG
Incidence of adverse events | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical Colledge, HUST, Wuhan, Hubei, China